CLINICAL TRIAL: NCT03808051
Title: Physiological-based Cord Clamping in Very Preterm Infants: a Multicentre Randomised Controlled Trial.
Brief Title: Aeration, Breathing, Clamping Study 3
Acronym: ABC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Medical Research Foundation, The Netherlands (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, PasABte, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL67770.058.18
Record Dates: First submitted 2019-01-01; First posted 2019-01-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Preterm Infant; Birth, Preterm
Keywords: Preterm infant; Cord clamping; Resuscitation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiological-based cord clamping (Experimental): Stabilisation of the infant is performed while the cord is intact and the cord will be clamped after the infant is cardiopulmonary stable. Stable is defined as the establishment of heart rate greater than 100 bpm and oxygen saturation above 85% while using supplemental oxygen lower than 40%. The maximum cord clamping time is 10 minutes and prior to cord clamping a trial of weaning from PPV to CPAP is performed. With the exception that the infant is stabilised close to the mother and the cord is clamped later, the infant will receive standard resuscitation interventions.
  Interventions: Procedure: Physiological-based cord clamping
- Time-based cord clamping (Active Comparator): Infants are clamped first and then moved to the standard resuscitation table for further treatment and intervention needed for cardiopulmonary stabilisation. Clamping is time based and performed immediately or delayed at 30-60 seconds, depending on the clinical condition of the infant. Uterotonic drugs are administered immediately after cord clamping.
  Interventions: Procedure: Time-based cord clamping

INTERVENTIONS:
Procedure: Physiological-based cord clamping — See Arm description.
  Arms: Physiological-based cord clamping
Procedure: Time-based cord clamping — See Arm description.
  Arms: Time-based cord clamping

SUMMARY:
Delayed cord clamping (DCC) in preterm infants results in a decrease in mortality and a trend towards fewer intraventricular haemorrhages. However, preterm infants needing immediate interventions for stabilisation or resuscitation were generally clamped immediately and excluded from trials, while these infants might benefit the most of DCC.

Studies in preterm lambs demonstrated that delaying cord clamping beyond ventilation onset resulted in more stable hemodynamic transition. This approach was called 'physiological-based cord clamping' (PBCC). The hypothesis of this study is that PBCC in preterm infants at birth will lead to an increase in intact survival when compared to standard care.

This study is a multicentre randomised controlled, parallel design, superiority trial, including preterm infants less than 30 weeks of gestation. The intervention is PBCC: stabilisation of the infant with the umbilical cord intact and only clamp the cord when the infant is stable. Stable is defined as the establishment of heart rate greater than 100 bpm and oxygen saturation above 85% while using supplemental oxygen lower than 40%. In the control group cord clamping will be performed time-based: infants are clamped first (at 30-60 seconds if the clinical condition allows) and then moved to the resuscitation table for further stabilisation.

The primary outcome will be intact survival at NICU discharge, defined as survival without cerebral injury (intraventricular haemorrhage ≥ grade 2 and/or periventricular leukomalacia ≥ grade 2 and/or periventricular venous infarction) and/or necrotizing enterocolitis (Bell stage ≥ 2).

ELIGIBILITY:
Inclusion Criteria:

* Infants born at a gestational age below 30 weeks in a participating centre.
* Parental consent (see 9.2).

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Significant congenital malformations influencing cardiopulmonary transition.
* Signs of acute placental abruption.
* Anterior placenta praevia or invasive placentation (accreta/percreta).
* Birth by emergency caesarean section (ordered to be executed within 15 minutes).
* Maternal general anaesthesia during caesarean section.
* Twin gestation with signs of Twin Transfusion Syndrome or Twin Anaemia Polycythemia Syndrome not treated with fetoscopic laser treatment.
* Multiple pregnancy > 2 (triplets or higher order).
* Decision documented to give palliative neonatal care.

In case of twin delivery by caesarean section it is not possible to perform PBCC in both infants. Both infants will be included: the first infant will receive standard treatment and the second infant will be randomised to either PBCC or standard treatment.

Max Age: 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 689 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Intact survival at NICU discharge | From date of randomization until the date of death or the date of NICU discharge, whichever came first, assessed up to 24 weeks.
  Intact survival is defined as survival without major cerebral injury (IVH ≥ grade 2 and/or PVL ≥ grade 2 and/or periventricular venous infarction) and/or NEC ≥ Bell stage 2.

SECONDARY OUTCOMES:
Rate of treatment failure | From birth until one hour of age.
  Treatment failure defined as the number of participants in which abortion of prescribed procedure (intervention or control) occurred and the reasons for abortion.
Short-term neonatal outcomes | From date of randomization until the date of death or the date of NICU discharge, whichever came first, assessed up to 24 weeks.
  Incidence of prematurity related morbidities during hospital stay.
Short-term maternal outcomes | From date of randomization until five days after intervention.
  Incidence of postpartum haemorrhage (> 1000 ml) and surgical site infection after caesarean section.
Neurodevelopmental outcome (Cognitive) at 2 years corrected age | Assesment at two years corrected age.
  Neurodevelopmental outcome assessed at 2 years corrected age by the standardized Bayley Scales of Infant Development III (BSID-III-NL), resulting in the Mental Developmental Index. A score of less than 85 (1 SD below the mean of 100) is considered as delayed development.
Neurodevelopmental outcome (Motor) at 2 years corrected age | Assesment at two years corrected age.
  Neurodevelopmental outcome assessed at 2 years corrected age by the standardized Bayley Scales of Infant Development III (BSID-III-NL), resulting in the Performance Developmental Index. A score of less than 85 (1 SD below the mean of 100) is considered as delayed development.
Functional outcome at 2 years corrected age | Assesment at two years corrected age.
  The proportion of participants with cerebral palsy, the proportion of participants with hearing loss requiring hearing aids and the proportion of participants with blindness.

OTHER OUTCOMES:
Parental perception and appreciation of stabilisation at birth | Sent within 1 week after birth.
  Questionnaire sent to parents concerning the perception and appreciation of the approach during birth and the perinatal stabilisation of the infant.

CONTACTS AND LOCATIONS:
Overall Officials: Arjan B Te Pas, Prof, Study Chair — Leiden University Medical Centre; Ronny Knol, MD, Principal Investigator — Erasmus Medical Centre Rotterdam
Locations (10):
- Netherlands (10):
  - Amsterdam University Medical Centre, location AMC, Amsterdam
  - Amsterdam University Medical Centre, location VU, Amsterdam
  - University Medical Centre Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Maastricht University Medical Centre, Maastricht
  - Radboud University Medical Centre, Nijmegen
  - Erasmus Medical Centre - Sophia Children's Hospital, Rotterdam
  - University Medical Centre Utrecht, Utrecht
  - Maxima Medical Centre, Veldhoven
  - Isala Clinics Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Knol R, Brouwer E, van den Akker T, DeKoninck PLJ, Onland W, Vermeulen MJ, de Boode WP, van Kaam AH, Lopriore E, Reiss IKM, Hutten GJ, Prins SA, Mulder EEM, d'Haens EJ, Hulzebos CV, Bouma HA, van Sambeeck SJ, Niemarkt HJ, van der Putten ME, Lebon T, Zonnenberg IA, Nuytemans DH, Willemsen SP, Polglase GR, Steggerda SJ, Hooper SB, Te Pas AB. Physiological versus time based cord clamping in very preterm infants (ABC3): a parallel-group, multicentre, randomised, controlled superiority trial. Lancet Reg Health Eur. 2024 Dec 4;48:101146. doi: 10.1016/j.lanepe.2024.101146. eCollection 2025 Jan. PMID 39717227
- [Derived] Willemsen SP, Knol R, Brouwer E, van den Akker T, DeKoninck PLJ, Lopriore E, Onland W, de Boode WP, van Kaam AH, Nuytemans DH, Reiss IKM, Hutten GJ, Prins SA, Mulder EEM, Hulzebos CV, van Sambeeck SJ, van der Putten ME, Zonnenberg IA, Te Pas AB, Vermeulen MJ. Physiological-based cord clamping in very preterm infants: the Aeration, Breathing, Clamping 3 (ABC3) trial-statistical analysis plan for a multicenter randomized controlled trial. Trials. 2024 Mar 4;25(1):164. doi: 10.1186/s13063-024-08014-y. PMID 38439024
- [Derived] Knol R, Brouwer E, van den Akker T, DeKoninck PLJ, Lopriore E, Onland W, Vermeulen MJ, van den Akker-van Marle ME, van Bodegom-Vos L, de Boode WP, van Kaam AH, Reiss IKM, Polglase GR, Hutten GJ, Prins SA, Mulder EEM, Hulzebos CV, van Sambeeck SJ, van der Putten ME, Zonnenberg IA, Hooper SB, Te Pas AB. Physiological-based cord clamping in very preterm infants: the Aeration, Breathing, Clamping 3 (ABC3) trial-study protocol for a multicentre randomised controlled trial. Trials. 2022 Oct 1;23(1):838. doi: 10.1186/s13063-022-06789-6. PMID 36183143